CLINICAL TRIAL: NCT05905094
Title: Effect of Postural Correction Exercise on Cervical Sagittal Posture, Proprioception, ROM and Head Flexion Angle in Forward Head Posture Among University Students.
Brief Title: Postural Correction Exercises Effect on Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/RCR&AHS/23/3003
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Musculoskeletal Disorder of the Neck

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postural correction exercises (Experimental): cervical retraction, shoulder shrugging, neck isometrics,
  Interventions: Other: Postural correction exercises

INTERVENTIONS:
Other: Postural correction exercises — Exercises to improve posture like shoulder shrugging, chin tuckin, neck isometrics

SUMMARY:
To determine the effect of postural correction exercise in universities students regarding cervical sagittal posture, head flexion angle in forward head posture.

DETAILED DESCRIPTION:
Informed consent will be taken from the participants, then we move further toward their demographics which will lead to initial readings after completion of authenticated questionnaire, then application of performing technique/exercise protocol by therapist and note the measurements again then interpret and analyze the data through data analyzing software which will lead to conclude the process.

ELIGIBILITY:
Inclusion Criteria:

* University students of age between 18 to 30 years.
* Smart devices addictions for one or more than one year and 2 h per day.
* CVA of less than 54°.
* Smartphone Addicted scale - short version SAS-SV

Exclusion Criteria:

* History of neurological symptoms and surgery to the neck and/or upper limbs.
* Smart devices usage less than one year.
* Unable to perform the exercises

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Smartphone Addicted scale - short version SAS-SV | 6 months
  It is used to measure smart phone addiction level. it is 10 items and self reported scale.
goniometery | 6 months
  to measure cervical range of motion of flexion, extension, side bending and rotation.
Cranio-vertebral angle | 6 months
  it is used to measure the degree of forward head posture. the angle will be less than 54 degree.

SECONDARY OUTCOMES:
Propioception | 6 months
  will be measure by laser point method in which sequence of movement will be performed. the deviation from normal pattern will be measure in CM and angle of deviation. there will be two reading one with eye open and 2nd with eye close.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- RIPHAH international university Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaghayegh Fard B, Ahmadi A, Maroufi N, Sarrafzadeh J. Evaluation of forward head posture in sitting and standing positions. Eur Spine J. 2016 Nov;25(11):3577-3582. doi: 10.1007/s00586-015-4254-x. Epub 2015 Oct 17. PMID 26476717
- [Background] Kim SY, Kim NS, Kim LJ. Effects of cervical sustained natural apophyseal glide on forward head posture and respiratory function. J Phys Ther Sci. 2015 Jun;27(6):1851-4. doi: 10.1589/jpts.27.1851. Epub 2015 Jun 30. PMID 26180334
- [Background] Sahrmann S, Azevedo DC, Dillen LV. Diagnosis and treatment of movement system impairment syndromes. Braz J Phys Ther. 2017 Nov-Dec;21(6):391-399. doi: 10.1016/j.bjpt.2017.08.001. Epub 2017 Sep 27. PMID 29097026